CLINICAL TRIAL: NCT04413396
Title: German Register of Outpatient Parenteral Antibiotic Therapy
Acronym: OPATReg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Clara Lehmann, Head of outpatient clinic, University of Cologne
Other Study IDs: OPATReg
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Implementation of OPAT in Germany

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatient parenteral antimicrobial therapy: Patients with an infectious disease that receive an outpatient parenteral antimicrobial therapy
  Interventions: Procedure: Outpatient Parenteral Antibiotic Therapy

INTERVENTIONS:
Procedure: Outpatient Parenteral Antibiotic Therapy — Application of outpatient parenteral antibiotic therapy in patients with infectious diseases to allow them to get discharged from hospital.

SUMMARY:
Many infectious diseases require a therapy that is administered intravenously due to a lack of oral treatments. Affected patients often have to stay weeks or even months in hospital just for receiving their therapy although they do not feel severely unwell.

Outpatient parenteral antibiotic therapy (OPAT) allows these patients under certain requirements to get discharged from hospital and apply the antibiotic treatment on their own. For these patients quality of life improves by feeling more comfortable at home and being able to participate in everyday life or even go back to work. For the hospitals a reduced inpatient health care means a clear reduction of costs.

The aim of OPATReg is to examine under which conditions the OPAT can be established at different locations of patient care. For this purpose, patients with APAT are to be treated and data collected at 7 university institutions in Germany. All centers have the expertise to provide comprehensive care for patients with infectious diseases, to transfer them from inpatient to outpatient care and to continue to provide care there.

If successful, the project should help to identify the potential of OPAT for all of Germany. If positive effects and feasibility can be demonstrated OPAT could become an important therapy option with many advantages for certain patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who get OPAT

Exclusion Criteria:

* patients who don't get OPAT

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults getting OPAT in one of the participating study sites
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with effective OPAT | 12 weeks
  Successful administration and completion of the antiinfective therapy
Number of Patients With Treatment-Related Adverse Events | 12 weeks
  side-effects of treatment and catheter-related infections
Number of Hospitals being able to apply OPAT | 12 weeks
  Feasibility of OPAT under differing hospital specific circumstances

CONTACTS AND LOCATIONS:
Overall Officials: Clara Lehmann, Prof., Study Chair — Head of Outpatient Department in ID, University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided